CLINICAL TRIAL: NCT06321393
Title: Effects of a Core Stabilization Exercise Program With the Abdominal drawing-in Maneuver Technique in Chronic Non-specific Low Back Pain With Lumbar Instability Using Telerehabilitation.
Brief Title: Effects of a CSE With ADIM in Chronic Non-specific Low Back Pain With Lumbar Instability Using Telerehabilitation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Torkamol Hunsawong, (PT, PhD), School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Thailand, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE662176
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain; Lumbar Instability
Keywords: Non-specific chronic low back pain with lumbar instability; lumbar instability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation-Based group (Experimental): A 7-week core stabilization exercise with abdominal drawing-in maneuver technique consist of 2 stages including the first stage (week 1-2) and the second stage (week 3-7) consisting of exercise program for 20-min sessions, with 3 sessions per week for 7 weeks. These exercise program will be provided to the participants via a weekly videocall with the main researcher as a telerehabilitation program.
  Interventions: Other: 7-week Core stabilization exercise with abdominal drawing-in maneuver technique
- Clinic-Based group (Active Comparator): The control group or clinic-base group will be provided the 7-week core stabilization exercise with abdominal drawing-in maneuver technique, the same as the experimental group, but control groups received the exercise program at the clinic according to the usual methods. At the first session of each week, an appointment will be set, and then the specific exercise for each week will be delivered and trained by the main researcher at the clinic. After completing weekly training, participants will perform their exercise routine as part of their daily home program.
  Interventions: Other: 7-week Core stabilization exercise with abdominal drawing-in maneuver technique

INTERVENTIONS:
Other: 7-week Core stabilization exercise with abdominal drawing-in maneuver technique — A 7-week core stabilization exercise with abdominal drawing-in maneuver technique consists of 2 stages, including the first stage (week 1-2) and the second stage (week 3-7) consisting of exercise program for 20-minute sessions with 3 sessions per week for 7 weeks. These exercise program will be provided to the participants via a weekly video call with the main researcher as a telerehabilitation program.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of telerehabilitation-based and clinic-based methods to deliver a Core Stabilization Exercise Program with the Abdominal Drawing-In Maneuver Technique (CSE with ADIM) on pain intensity, functional ability, quality of life, and satisfaction in chronic low back pain patients with lumbar instability.

The main question it aims to answer is: Is there a difference between the effectiveness of telerehabilitation-based and clinic-based CSE with ADIM on pain intensity, functional ability, quality of life, and satisfaction in chronic low back pain patients with lumbar instability?

Participants will perform a 7-week core stabilization exercise with the abdominal drawing-in maneuver technique, consisting of an exercise program for 20-minute sessions with 3 sessions per week. These exercise programs will be provided to the participants via a weekly video call with the main researcher as a telerehabilitation program. At the first session of each week, the researcher will provide supervision via video call with the participant for the exercise program. The participants will perform the exercise by following the video demonstration. After completing weekly training, participants will perform their exercise routine as part of their daily home program.

If there is a comparison group: researchers will compare The control group (clinical-base group) will be provided the 7-week core stabilization exercise with abdominal drawing-in maneuver technique, the same as the experimental group, but control groups received the exercise program at the clinic according to the usual methods. At the first session of each week, an appointment will be set, and then the specific exercise for each week will be delivered and trained by the main researcher at the clinic. After completing weekly training, participants will perform their exercise routine as part of their daily home program to see if there are any differences in pain intensity, functional ability, quality of life, and satisfaction in chronic low back pain patients with lumbar instability between the experimental and control groups.

DETAILED DESCRIPTION:
This study is conducted as a single-blinded, randomized control trial to compare the effectiveness of telerehabilitation-based and clinic-based methods to deliver CSE with ADIM on pain intensity, functional ability, quality of life, and satisfaction in chronic low back pain patients with lumbar instability. Participants will be non-specific chronic low back pain patients with lumbar instability, which will be screened by history and physical examination. Lumbar instability will be diagnosed using the Screening Tool for Patients with Lumbar Instability Questionnaire, 14 items were yes-or-no questions. If "yes" answers are more than 6/14, this score represents lumbar instability and will be diagnosed by special tests with at least two positive signs from three special tests consisting of: 1) Painful catch sign; 2) Aberrant movement sign; and 3) Prone instability test.

The estimation of the sample is based on a previous study of Chalermsan et al. (2016. Based on this study, a standard deviation of pain intensity after treatment for both groups were used to calculate the sample size for a power of 80% at 5% significance, and a dropout rate of 30% allowed for estimating the final sample. Therefore, the sample size will be 15 participants per group, and the total number of participants will be 30. The allocation sequence will be generated using the random number function in Excel. All participants will be randomly allocated to either the telerehabilitation-based group or the clinic-based group using stratified random allocation by age groups and gender.

The data collection process in this study. After participants receive a screen test and sign the informed consent form, a baseline assessment will be conducted by the assessor before randomization. The outcome measurement includes pain level assessment using the numerical rating scale (NRS), participation restriction using the Oswestry disability index (ODI), activity limitation using the Roland Morris Disability Questionnaire (RMDQ), quality of life using the 36-item Short Form Survey (SF-36), and lumbar joint repositioning sense to measure proprioception. Regarding lumbar joint repositioning sense measurement, participants will be asked to sit with their hips and knees at 90 degrees, feet supported, and arms resting on their thighs. The assessor will guide the participant's lumbar spine into a mid-range position between a posterior and anterior pelvic tilt. The assessor then uses a 10-centimeter tape measure on the participant's lumbar, with the center of the tape marking sacral segment 1 (S1) as the measurement start point. A laser pointer placed on a stable base and adjusted to be level is in a in a position to have the mark line directly on the start point. The participant will be instructed to remember this position before moving the pelvis twice from maximum anterior to maximum posterior tilt for approximately five seconds before returning to neutral position. The distance from the starting point will be measured in centimeters using the laser line on the tape measure. This protocol will be conducted by an assessor (researcher number 1) who is a licensed physical therapist and blinded to group allocation. Then participants will be randomly allocated into one of two groups in this study: either the telerehabilitation-based group or the clinic-based group, by the assistant researcher. All outcome measures will be reassessed after completing the seven-week intervention. Furthermore, a satisfaction questionnaire will be used to determine satisfaction, and then the satisfaction of participants will be determined using a 5-point Likert scale questionnaire.

The intervention of this study is a 7-week core stabilization exercise with abdominal drawing-in maneuver technique, or CSE with ADIM. All participants received a 7-week CSE with ADIM. However, the method of receiving the exercise program in the experimental group (telerehabilitation-based group) will be telerehabilitation via video call with the main researcher. At the first session of each week, the researcher will provide supervision via video call with the participant for the exercise program. The participants will perform the exercise by following the video demonstration. In this session, the main researcher will supervise the participants as they do the exercise. The session will start with the participant and the main researcher watching the video demonstrating the exercise program together. After watching the video, the participants can ask a question in case they have any doubts about how to do the exercise. Then the participants will be asked to perform the exercise, and the main researcher will observe and advise or correct in case the participant cannot perform the exercise correctly. For the rest of the week, the participants will perform the exercise by themselves. In case they want to ask any questions, they can contact the main researcher via line application. In the control group (clinic-based group), at the first session of each week, an appointment with the main researcher will be set, and then the specific exercise for each week will be delivered and trained by the main researcher at the clinic. After completing weekly training, participants will perform their exercise routine as part of a daily home program.

The statistical analysis will be performed using SPSS version 22.0 for Windows (IBM Corporation, Armonk, NY, USA). The Shapiro-Wilk test will be used to test the normality of the data. All data analysis will be performed with an intention-to-treat analysis. The data will be presented as means, standard deviations (SD), 95% CI, percentage, ratio, or mode, and interquartile as appropriate. The analysis of comparisons within the pre- and post-intervention in each group will use a pair T-test. The analysis of comparative data between the telerehabilitation-based group and the clinic-based group will use an analysis of covariance (ANCOVA). Because the randomization process does not ensure that the groups have identical baseline characteristics, the researchers conducted an ANCOVA to compare the differences in outcome measures between the groups. In this analysis, the pre-test scores of each outcome will be used as a covariate to estimate the adjusted mean differences and 95% confidence intervals for each outcome measure in each group. The researcher will interpret Partial Eta Squared effect sizes as either large (≥ 0.80), medium (0.50-0.79), or small (0.20-0.49) (Richardson et al., 2011), and the level of significance will be set at a p-value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females.
2. Aged between 18 - 60 years old.
3. Onset of back pain lasting more than 12 weeks.
4. Lumbar instability will be diagnosed using a score of at least 6 out of 14 on the Screening Tool for Patients with Lumbar Instability Questionnaire in Thai version.
5. Presented at least two positive signs from three special tests of the following provocation tests: Painful catch, aberrant movement sign, or prone instability test.
6. Pain intensity at rest has a pain level with a numerical rating scale (0-10 NRS) 3-7/10 points.
7. Never receive the treatment by core stabilization exercise during 3 months before participate in this study.
8. Participants must have a smart phone, tablet, or other electronic device with a camera and install the line application on the device. They can perform the basic operations of these devices by themselves.
9. Participants have the ability to read and write Thai fluently.

Exclusion Criteria:

1. Onset of serious spinal pathology: spinal fracture, spinal malignancy, or spinal infection.
2. Have been diagnosed with osteoporosis, ankylosing spondylitis, or spondyloarthritis.
3. History of spinal surgery and/or lower extremity.
4. Cauda equina syndrome.
5. Presented at least 2 out of 3 signs of neurological deficit including reflex abnormality or loss of sensation of lower limbs associated with the spinal nerve root and weakness of lower limbs (muscle power less than grade 3 using manual muscle test) (Macedo et al., 2008).
6. Pregnancy or during breast feeding.
7. Body mass index (BMI) > 30 kg/m2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
11-ponits Numerical Rating Scale (0-10 NRS) | Baseline and after Week 7
  The 11-point numerical rating scale (0-10 NRS) will be used to assess low back pain intensity at rest. The NRS consists of a line or box scale with numbers in descending order, where 0 represents no pain and 10 represents the worst imaginable pain.

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | Baseline and after Week 7
  Oswestry disability index (ODI) will be used to assess physical disability in patients with low back pain to determine participation restrictions. The ODI consists of 10 patient-completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability ) to 100% (most severe disability).
Roland Morris Disability Questionnaire (RMDQ) | Baseline and after Week 7
  Roland Morris Disability Questionnaire (RMDQ) will be used to assess physical disability in patients with low back pain to determine activity limitations. The RMDQ consists of 24 items with a yes or no answer. The possible total score can be 0 to 24, with 0 interpreted as no disability and 24 interpreted as maximum disability.
36-item Short Form Survey (SF-36) | Baseline and after Week 7
  The 36-item Short Form Survey (SF-36) will be used to assess quality of life. The SF-36 contains 36 health-related questions divided into eight domains including 1) physical function, 10 items; 2) role limited by physical problem, 4 items; 3) bodily pain, 2 items; 4) general health, 6 items; 5) vitality, 4 items; 6) social-functioning, 2 items; 7) role limited by emotional problem, 3 items; 8) mental health, 5 items; each with a choice of a Likert-type scale. The total possible score can be 0 to 100 (a high scores represents a good quality of life).
Lumbar joint reposition sense error | Baseline and after Week 7
  Lumbar joint reposition sense error will be used to assess proprioception sense in the lumbar spine. The distance from the starting point will be measured in centimeters using the laser line on the tape measure. This examination will be carried out three times with one-minute rest intervals and the average values of the measurements that will be taken into consideration for the analysis. If the distance from the starting point is large, it means that the proprioceptive sense of the lower back is worse.
Satisfaction questionnaire | After Week 7
  Satisfaction questionnaire consisting of five aspects such as program usability, media, teleconsultation, researcher's response to participant suggestions. The total scores will be divided by 25 and multiplied by 100 to derive a percentage. Higher scores indicate greater satisfaction levels, whereas lower scores indicate lower levels of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chutimon Kongsa, Study Chair — Physical therapy Unit, Suddhavej Hospital, Faculty of Medicine, Mahasarakham UniversityMa
Locations (1):
- Miss Chutimon Kongsa, Maha Sarakham, Mahasarakham, Thailand